CLINICAL TRIAL: NCT02895594
Title: Outcome of Surgery for Idiopathic Macular Holes
Acronym: TROMAC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_YLR_2015_1
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Idiopathic Macular Hole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Retrospective medical chart review of patients undergoing surgical repair of idiopathic macular hole

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from primary idiopathic macular hole and treated by retinal repair surgery

Exclusion Criteria:

* Presence of other retinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by retinal repair surgery for idiopathic macular hole
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Primary closure of macular hole after repair surgery | within six months after surgery